CLINICAL TRIAL: NCT02972892
Title: Multi-site Anesthesia Randomized Controlled STudy of End Tidal Control (Et Control) Compared to Conventional Anesthesia Results (MASTER-Anesthesia Trial)
Brief Title: Multi-site Anesthesia Randomized Controlled STudy of End Tidal Control Compared to Conventional Anesthesia Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 123.07-2015-GES-0002
Record Dates: First submitted 2016-11-14; First posted 2016-11-25 (Estimated); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Et Control Performance in Adult Population Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Et Control (Experimental): Subjects, meeting the American Society of Anesthesiologists status classification system 1-3, to undergo a surgical procedure with inhaled anesthesia using the investigational Et Control option intervention. For Subjects under the Et Control option, the investigator will use and initiate Et Control after the airway is secured and mechanical ventilation is initiated. Machine log data is collected when the investigator initiates the start of anesthesia case on the Aisys CS2. Adjustments to the anesthesia machine settings, discontinuation of use of the investigational Et Control option, and changes to treatment are based upon clinician judgment for the well being of the subject.
  Interventions: Device: Et Control Feature
- Control Arm (Active Comparator): Subjects, meeting the American Society of Anesthesiologists status classification system 1-3, to undergo a surgical procedure with inhaled anesthesia using conventional fresh gas intervention. For subjects under the conventional option, the investigator will use their conventional means to adjust the vaporizer and mixer, and monitor the patient gas concentrations with the legally marketed Aisys CS2 anesthesia machine without the investigational Et Control feature.
  Interventions: Device: Conventional Fresh Gas

INTERVENTIONS:
Device: Et Control Feature — Subjects using Et Control option; the investigator will use and initiate Et Control after the airway is secured and mechanical ventilation is initiated. Machine log data is collected when the investigator initiates the start of anesthesia case on the Aisys CS2. Adjustments to the anesthesia machine settings, discontinuation of use of the investigational Et Control option, and changes to treatment are based upon clinician judgment for the wellbeing of the subject. The clinician must continuously monitor measured inspired and end tidal oxygen and anesthetic concentrations to assess individual responses and compare to the target concentrations.
  Arms: Et Control
Device: Conventional Fresh Gas — Subjects to undergo a surgical procedure with inhaled anesthesia meeting the American Society of Anesthesiologists status classification system 1-3. Subjects using conventional option; the investigator will use their conventional means to adjust the vaporizer and mixer, and monitor the patient gas concentrations with the legally marketed Aisys CS2 anesthesia machine without the investigational Et Control feature. Machine log data collection will end, when an "end case" is confirmed on the Aisys CS2 at the end of the anesthesia case.
  Arms: Control Arm

SUMMARY:
This is a clinical, single blind, randomized, prospective research study. The purpose of this pivotal study is to collect and analyze data on the investigational End tidal Control (Et Control) option feature. To demonstrate that End tidal Control (Et Control) performance is non-inferior to conventional anesthesia practice in an adult surgery population by comparing the performance of the Et Control Arm (investigational arm) to the Control Arm (fresh gas mode).

DETAILED DESCRIPTION:
The purpose of this pivotal study is to demonstrate that End tidal Control performance is non-inferior to conventional anesthesia practice in an adult surgery population, and support a marketing application in the U.S. for clearance of this feature.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years old or greater.
2. Scheduled to undergo general inhaled anesthesia that can be safely exposed to 100% oxygen for up to 2 minutes during general anesthesia.
3. Expected to have airway secured with laryngeal mask airway (LMA) or endotracheal tube.
4. Undergoing a surgical procedure that is anticipated by the investigator to take greater than or equal to 1 hour (operative time measured from induction to cessation of general inhalation anesthetic).
5. American Society of Anesthesiologists (ASA) status classification system I through III:

   1. ASA Physical Status 1 = a normal healthy patient
   2. ASA Physical Status 2 = a patient with mild systemic disease
   3. ASA Physical Status 3 = a patient with severe systemic disease
6. Undergoing intravenous induction.
7. Ability to provide written informed consent.

Exclusion Criteria:

1. Have emergency medical condition requiring surgery.
2. Are female subjects, who are pregnant or lactating.
3. Any subject undergoing cardiac bypass surgery.
4. Any subject undergoing open chest surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Seering, MD, Principal Investigator — University of Iowa Healthcare
Locations (4):
- United States (4):
  - Loma Linda University, Loma Linda, California
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa Healthcare, Iowa City, Iowa
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared and reviewed are: adverse events listing, serious adverse event (SAE)/unanticipated adverse device effects (UADE) summary, demographics, surgical procedure, treatment allocation, early termination, critical protocol deviations, device malfunction reports, and plotted data (Et Control subjects with adverse events only). These items are listed in the Data Safety Monitoring Board (DSMB) Charter.
Supporting Information: Study Protocol
Time Frame: Data will be available according to the following timeline: (1) when a minimum of 20 Et Control subjects enrolled and at least 2 sites initiated and enrolling; (2) 50% enrollment; (3) 80% enrollment; and (4) 100% enrollment.
Access Criteria: Members of the DSMB will have access to the data listed under the Plan Description section. Reports will consist of tables, listings, and figures; and will be delivered electronically at least 7 calendar days prior to the date of each DSMB meeting.

REFERENCES:
- [Derived] McCabe MD, Dear GL, Klopman MA, Garg K, Seering MS. End-Tidal Control Versus Manual Control of Inhalational Anesthesia Delivery: A Randomized Controlled Noninferiority Trial. Anesth Analg. 2024 Oct 1;139(4):812-820. doi: 10.1213/ANE.0000000000007132. Epub 2024 Jul 19. PMID 39028663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in June 2017 and was completed in July 2018. 248 subjects were enrolled at 4 sites. Males and females,18 years or older and scheduled to undergo general inhaled anesthesia during surgery, were screened for enrollment into this study. Subjects enrolled were randomized at a 1:1 ratio to either the Et Control Arm or the Control Arm. Randomization was stratified based on the Investigator, subject's pre-existing hypertension status, and subject's ASA status classification.
Pre-assignment Details: Subjects are considered enrolled at the time of informed consent. After consent, subjects were screened against the inclusion/exclusion criteria according to standard procedures of the investigational site.
Period: Overall Study
Arm/Group | Et Control | Control Arm
Started | 110 | 118
Completed | 101 | 116
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat population included all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Et Control | Control Arm | Total
Number analyzed (Participants) | 110 | 118 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 91 | 181
  >=65 years | 20 | 27 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 63 | 114
  Male | 59 | 55 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 98 | 105 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 21 | 20 | 41
  White | 77 | 81 | 158
  More than one race | NA — Not an option on the CRF | NA — Not an option on the CRF | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 110 | 118 | 228

OUTCOME MEASURES:

1. Primary Outcome: Percent Duration Without Large Deviation of End-Tidal Anesthetic Agent (EtAA) Based on Extraction Algorithm (ALG)
Description: Percent duration of EtAA concentration during steady state maintained within the acceptable limit, which is defined as the greater of 5% of the steady state inhaled anesthetic agent concentration and 0.6% v/v for Desflurane (Des), 0.2% v/v for Sevoflurane (Sev), or 0.1% v/v for Isoflurane (Iso). The percent duration is the weighted average of all steady states for a subject, using the duration of steady state as the weight. Steady state concentration is based on an extraction algorithm described in Appendix 2 of the protocol.
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent duration
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
percent duration | 91.7 (10.82) | 80.8 (17.93)
Statistical Analysis 1: Comparison: Et Control vs Control Arm; Using t-test, comparison of the weighted average percent duration between the Et Control and control device was performed by calculating the difference and its 95% 2-sided confidence interval between the two arms. Non-inferiority will be concluded if the lower limit of the 95% confidence interval is ≥ -5% for both EtAA; Test type: Non-Inferiority — Using t-test, comparison of the weighted average percent duration between the Et Control and control device was performed by calculating the difference and its 95% 2-sided confidence interval between the two arms. Non-inferiority will be concluded if the lower limit of the 95% confidence interval is ≥ -5% for both EtAA; p < .001, t-test, 2 sided; Mean Difference (Net) = 10.9, 95% CI 2-sided [6.89 to 15.01]

2. Primary Outcome: Percent Duration Without Large Deviation of EtAA Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Percent duration of EtAA concentration during steady state maintained within the acceptable limit, which is defined as the greater of 5% of the steady state inhaled anesthetic agent concentration and 0.6% v/v for Desflurane (Des), 0.2% v/v for Sevoflurane (Sev), or 0.1% v/v for Isoflurane (Iso). The percent duration is the weighted average of all steady states for a subject, using the duration of steady state as the weight. Data obtained using the clinicians' or Investigators' recorded target (TGT) values of anesthetic agent and oxygen for the Control Arm and using the set target values for the Et Control Arm.
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent duration
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
percent duration | 98.0 (2.05) | 45.9 (31.45)
Statistical Analysis 1: Comparison: Et Control vs Control Arm; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < .001, t-test, 2 sided; Mean Difference (Net) = 52.1, 95% CI 2-sided [46.25 to 57.95]

3. Primary Outcome: Percent Duration Without Large Deviation of End-Tidal Oxygen (EtO2) Based on Extraction Algorithm (ALG)
Description: Percent duration of EtAA concentration during steady state maintained within the acceptable limit, which is defined as the greater of 5% of the steady state inhaled anesthetic agent concentration and 0.6% v/v for Desflurane (Des), 0.2% v/v for Sevoflurane (Sev), or 0.1% v/v for Isoflurane (Iso). The percent duration is the weighted average of all steady states for a subject, using the duration of steady state as the weight. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent duration
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
percent duration | 98.1 (2.76) | 92.8 (14.38)
Statistical Analysis 1: Comparison: Et Control vs Control Arm; Using t-test, comparison of the weighted average percent duration between the Et Control and control device will be performed by calculating the difference and its 95% 2-sided confidence interval between the two arms. Non-inferiority will be concluded if the lower limit of the 95% confidence interval is ≥ -5% for EtO2; Test type: Non-Inferiority — Using t-test, comparison of the weighted average percent duration between the Et Control and control device will be performed by calculating the difference and its 95% 2-sided confidence interval between the two arms. Non-inferiority will be concluded if the lower limit of the 95% confidence interval is ≥ -5% for EtO2; p < .001, t-test, 2 sided; Mean Difference (Net) = 5.3, 95% CI 2-sided [2.64 to 8.04]

4. Primary Outcome: Percent Duration Without Large Deviation of EtO2 Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Percent duration of EtAA concentration during steady state maintained within the acceptable limit, which is defined as the greater of 5% of the steady state inhaled anesthetic agent concentration and 0.6% v/v for Desflurane (Des), 0.2% v/v for Sevoflurane (Sev), or 0.1% v/v for Isoflurane (Iso). The percent duration is the weighted average of all steady states for a subject, using the duration of steady state as the weight. Values based on clinicians' or Investigators' recorded target values (TGT)
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent duration
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
percent duration | 98.8 (1.49) | 41.0 (40.65)
Statistical Analysis 1: Comparison: Et Control vs Control Arm; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p < .001, t-test, 2 sided; Mean Difference (Net) = 44.5, 95% CI 2-sided [35.56 to 53.41]

5. Secondary Outcome: Efficacy Response Time EtAA Based on Extraction Algorithm (ALG)
Description: Response time: time to reach 90% of the desired change in EtAA steady state mean concentration. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 283 | 184
Seconds | 73 (174.1) | 196 (378.3)

6. Secondary Outcome: Efficacy: Response Time for EtAA Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: time to reach 90% of the desired change in EtAA and EtO2 steady state mean concentration. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 520 | 281
Seconds | 23 (40.9) | 196 (455.0)

7. Secondary Outcome: Efficacy Response Time for EtO2 Based on Extraction Algorithm (ALG)
Description: Response time: time to reach 90% of the desired change in EtO2 steady state mean concentration. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes.
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 238 | 318
Seconds | 93 (77.3) | 246 (346.8)

8. Secondary Outcome: Efficacy: Response Time for EtO2 Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Response time: time to reach 90% of the desired change in EtAA and EtO2 steady state mean concentration. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 240 | 209
Seconds | 129 (451.7) | 406 (727.8)

9. Secondary Outcome: Efficacy: Settling Time for EtAA Based on the Extraction Algorithm (ALG)
Description: Settling time: time to achieve the desired EtAA steady state mean concentration. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 283 | 184
Seconds | 105 (181.9) | 165 (186.4)

10. Secondary Outcome: Efficacy: Settling Time for EtAA Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Settling time: time to achieve the desired EtAA steady state mean concentration. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 520 | 281
Seconds | 23 (40.9) | 196 (455.0)

11. Secondary Outcome: Efficacy: Settling Time for EtO2 Based on the Extraction Algorithm (ALG)
Description: Settling time: time to achieve the desired EtO2 steady state mean concentration. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 238 | 318
Seconds | 123 (117.5) | 235 (213.2)

12. Secondary Outcome: Efficacy: Settling Time for EtO2 Based on Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: time to achieve the desired EtO2 steady state mean concentration. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 240 | 209
Seconds | 167 (121.1) | 815 (1327.2)

13. Secondary Outcome: Efficacy: Overshoot Amount of the Desired EtAA Based on Extraction Algorithm (ALG)
Description: Overshoot amount of the desired EtAA from steady state mean concentration. Command Overshoot is defined as the maximum value beyond the desired end tidal concentration from the start of the step change until the Settling Time. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent to mean
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 283 | 184
percent to mean | 8.85 (12.026) | 6.54 (13.576)

14. Secondary Outcome: Efficacy: Overshoot Amount of the Desired EtAA Amount Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Overshoot amount of the desired EtAA from steady state mean concentration. Command Overshoot is defined as the maximum value beyond the desired end tidal concentration from the start of the step change until the Settling Time. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent to mean
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 519 | 278
percent to mean | 5.28 (6.953) | 12.09 (27.085)

15. Secondary Outcome: Efficacy: Overshoot Amount of Desired EtO2 Amount Based on the Extraction Algorithm (ALG)
Description: Overshoot amount of the desired EtO2 from steady state mean concentration. Command Overshoot is defined as the maximum value beyond the desired end tidal concentration from the start of the step change until the Settling Time. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent to mean
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 238 | 318
percent to mean | 3.47 (8.238) | 2.80 (11.373)

16. Secondary Outcome: Efficacy: Overshoot Amount of Desired EtO2 Amount Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Overshoot amount of the desired EtO2 from steady state mean concentration. Command Overshoot is defined as the maximum value beyond the desired end tidal concentration from the start of the step change until the Settling Time. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of each steady state, an average of approximately 60 minutes
Population: Intent-to-treat population includes all randomized subjects
Measure: Mean (Standard Deviation); unit: percent to mean
Units Other Than Participants: steady states
Arm/Group | Et Control | Control Arm
Number analyzed (Participants) | 110 | 118
Number analyzed (steady states) | 240 | 209
percent to mean | 2.14 (6.277) | 11.13 (20.662)

17. Secondary Outcome: Accuracy of Et Control in Maintaining EtAA Control Between User Set Target and Settling End Tidal Concentrations Based on the Extraction Algorithm (ALG)
Description: Accuracy of Et Control in maintaining EtAA control between user set target and settling end tidal concentrations. Calculated for Et Control arm only. The accuracy measures include absolute difference between steady state and set EtAA concentrations. The acceptable limits defined by the primary endpoint were: 0.1% of Isoflurane, 0.2% for Sevoflurane, 0.6% for Desflurane. As a measure of Absolute Difference between Steady State and Set EtAA Concentration (%). Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of surgery, average of 112.1 minutes (+/- 78.7 minutes)
Population: Subjects randomized to the ET control arm of the study who underwent surgery
Measure: Mean (Standard Deviation); unit: Absolute Difference (%)
Units Other Than Participants: steady states
Groups:
- ET Control - Desflurane: Subjects randomized to the ET Control arm of the trial who received Desflurane as their inhaled anesthetic agent.
- Et Control - Isoflurane: Subjects randomized to the ET Control arm of the trial who received Isoflurane as their inhaled anesthetic agent.
- ET Control - Sevoflurane: Subjects randomized to the ET Control arm of the trial who received Sevoflurane as their inhaled anesthetic agent.
- ET Control - All: Summary of all Subjects randomized to the ET Control arm of the trial combining all anesthetic agents.
Arm/Group | ET Control - Desflurane | Et Control - Isoflurane | ET Control - Sevoflurane | ET Control - All
Number analyzed (Participants) | 27 | 17 | 56 | 100
Number analyzed (steady states) | 50 | 54 | 178 | 282
Absolute Difference (%) | 0.11 (0.056) | 0.04 (0.031) | 0.04 (0.026) | 0.05 (0.043)

18. Secondary Outcome: Accuracy of ET Control in Maintaining EtAA Control Between User Set Target and Settling End Tidal Concentrations Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Accuracy of ET Control in maintatining EtAA between user set target and settling end tidal concentrations. Calculated for ET Control arm only. The accuracy measures include absolute difference between steady state and set EtAA concentrations. The acceptable limits defined by the primary endpoint were: 0.1% of Isoflurane, 0.2% for Sevoflurane, 0.6% for Desflurane. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of Surgery
Population: Subjects Randomized to the ET control arm of the study who underwent surgery
Measure: Mean (Standard Deviation); unit: Absolute Difference (%)
Units Other Than Participants: steady states
Arm/Group | ET Control - Desflurane | Et Control - Isoflurane | ET Control - Sevoflurane | ET Control - All
Number analyzed (Participants) | 27 | 17 | 56 | 100
Number analyzed (steady states) | 85 | 72 | 362 | 519
Absolute Difference (%) | 0.10 (0.054) | 0.03 (0.031) | 0.04 (0.027) | 0.05 (0.04)

19. Secondary Outcome: Accuracy of Et Control in Maintaining EtO2 Between User Set Target and Settling End Tidal Concentrations Based on the Extraction Algorithm (ALG)
Description: Accuracy of Et Control in maintaining EtO2 control between user set target and settling end tidal concentrations. Calculated for Et Control arm only. outcome measures the absolute difference between Steady State and Set EtO2 Concentrations. The acceptable limit defined by the primary endpoint was < 5% v/v. Values based on the extraction algorithm described in Appendix 2 of the protocol (ALG).
Time Frame: Duration of surgery, average of 112.1 minutes (+/- 78.7 minutes)
Population: Subjects randomized to the ET control arm of the study who underwent surgery.
Measure: Mean (Standard Deviation); unit: Absolute Difference (%)
Units Other Than Participants: steady states
Arm/Group | ET Control - Desflurane | Et Control - Isoflurane | ET Control - Sevoflurane | ET Control - All
Number analyzed (Participants) | 27 | 17 | 56 | 100
Number analyzed (steady states) | 58 | 34 | 146 | 238
Absolute Difference (%) | 0.57 (0.594) | 0.62 (0.613) | 0.64 (0.932) | 0.62 (0.818)

20. Secondary Outcome: Accuracy of Et Control in Maintaining EtO2 Between User Set Target and Settling End Tidal Concentrations Based on Clinician's or Investigators' Recorded Target Values of Anesthetic Agent and Oxygen (TGT)
Description: Accuracy of Et Control in maintaining EtO2 control between user set target and settling end tidal concentrations. Calculated for Et Control arm only. outcome measures the absolute difference between Steady State and Set EtO2 Concentrations. The acceptable limit defined by the primary endpoint was < 5% v/v. Values based on clinicians' or Investigators' recorded values (TGT).
Time Frame: Duration of surgery, average of 112.1 minutes (+/- 78.7 minutes)
Population: Subjects randomized to the ET control arm of the study who underwent surgery
Measure: Mean (Standard Deviation); unit: Absolute Difference (%)
Units Other Than Participants: steady states
Arm/Group | ET Control - Desflurane | Et Control - Isoflurane | ET Control - Sevoflurane | ET Control - All
Number analyzed (Participants) | 27 | 17 | 56 | 100
Number analyzed (steady states) | 60 | 33 | 147 | 240
Absolute Difference (%) | 0.62 (0.632) | 0.61 (0.585) | 0.64 (0.863) | 0.63 (0.774)

21. Other Pre Specified Outcome: Inhaled Anesthetic Agent
Description: Usage of inhaled anesthetic agent
Time Frame: Duration of Procedure
Reporting Status: Not Posted

22. Other Pre Specified Outcome: User Interactions
Description: Number of user interactions
Time Frame: Duration of Procedure
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Discharge From the Operating Room
Description: Time to discharge from the operating room
Time Frame: End of surgery to time of last breath
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse even assessment was conducted from the time the subject provided consent to the end of the subject's participation in the study. Approximately 30 hours
Description: For each Adverse Event, the following information was recorded: Description of AE, Onset date/time, relationship to device/study, relationship to anesthetic agent, relationship to surgical procedure, resolution, anticipated/unanticipated, serious AE, outcome, severity, and treatment given.
Arm/Group | Et Control | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/116
Serious Adverse Events (participants affected / at risk) | 1/104 | 1/116
Other Adverse Events (participants affected / at risk) | 36/104 | 43/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Et Control (N=104) | Control Arm (N=116)
Bile Leak (Hepatobiliary disorders) | 0 (0) | 1 (1)
Vision Loss (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Et Control (N=104) | Control Arm (N=116)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bladder Spasms (Renal and urinary disorders) | 1 (1) | 0 (0)
Post-Operative Pain (Surgical and medical procedures) | 1 (1) | 1 (1)
Inadvertent Cystotomy and Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Post Operative Pain of 10 (Surgical and medical procedures) | 0 (0) | 1 (1)
Intraoperative Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0)
Intractable Pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Pain 7 out of 10 (Surgical and medical procedures) | 2 (2) | 2 (2)
Elevated Heart Rate and Breathing (Surgical and medical procedures) | 0 (0) | 1 (1) — Trouble breathing and inadequate reversal of neuromuscular blocking agent led to elevated heart rate and elevated blood pressure which was resolved by sugammadex
Bladder Wall Damage (Renal and urinary disorders) | 1 (1) | 0 (0)
Left Thigh Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain 8 of 10 (Surgical and medical procedures) | 2 (2) | 3 (3)
Hypotension (general) (Vascular disorders) | 3 (3) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
NIBP SBP>160 mmHg for >5 min (Vascular disorders) | 15 (15) | 24 (24)
NIBP MAP >120 mmHg for > 5 min (Vascular disorders) | 5 (5) | 5 (5)
HR <45bpm more than 5 min (Cardiac disorders) | 2 (2) | 0 (0)
Emergence Delay (Surgical and medical procedures) | 1 (1) | 0 (0)
Throat Pain (General disorders) | 0 (0) | 1 (1)
Oral Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Pain 9 of 10 (Surgical and medical procedures) | 1 (1) | 1 (1)
Intermittent Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0)
Dizziness, photophobia, and delay in discharge from PACU (Surgical and medical procedures) | 0 (0) | 1 (1)
Low Urine Output (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Large Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SpO2 < 90% for more than 5 min (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Severe Post Operative Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
HR >110bpm more than 5 min (Cardiac disorders) | 7 (7) | 5 (5)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NIPB MAP <55 mmHg for >5 min (Vascular disorders) | 3 (3) | 1 (1)
NIBP SBP <70 mmHg for >5 min (Vascular disorders) | 2 (2) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Corneal Abrasion (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02972892/Prot_SAP_000.pdf